CLINICAL TRIAL: NCT01924793
Title: An Open Label Study to Examine the Effects of DAS181 Administered by Dry Powder Inhaler (DPI) or Nebulized Formulation in Immunocompromised Subjects With Parainfluenza (PIV) Infection
Acronym: PIV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ansun Biopharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAS181-2-06
Record Dates: First submitted 2013-07-11; First posted 2013-08-19 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Parainfluenza
MeSH Terms: conditions — Paramyxoviridae Infections | interventions — Dietary Fiber

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Formulation of DAS181-F02 Dry Powder in Bulk (Experimental): The DAS181-F02 nebulized formulation includes 10mL of normal saline to prepare a liquid solution referred to as DAS181-F02 nebulized.
  Dry Powder Inhaled Dose:
  Non-ventilated subjects, capable of using a cyclohaler, will be treated by Dry Powder Inhalation. Each subject will receive a targeted daily dose of 10mg for 7 days for a total of 70mg of DAS181-F02. If a subject requires ventilation, the subject will be allowed to continue dosing following the Nebulized formulation instruction.
  Interventions: Drug: DAS181-F02 Dry Powder in Bulk
- Nebulized Formulation Inhaled Dose (Experimental): Subjects unable to use the Dry Powder Inhaler (as determined by site Investigator) on continuous positive airway pressure (CPAP), Bi-level positive airway pressure (BIPAP) or requiring mechanical ventilation will be treated by Nebulized formulation. The subject will remain on the nebulized formulation for the duration of the study regardless of ventilation status. DAS-F02 10 mg will be utilized to prepare the nebulized solution per the Study Reference Manual.
  Multiple methods (T piece, face mask, direct to ET tube) will be allowed for the nebulized dose administration. Detailed specification for nebulized dose administration will be defined in the Study Reference Manual.
  Interventions: Drug: DAS181-F02 Nebulized Formulation Inhaled Dose

INTERVENTIONS:
Drug: DAS181-F02 Dry Powder in Bulk — Administered via DPI
  Arms: Formulation of DAS181-F02 Dry Powder in Bulk
Drug: DAS181-F02 Nebulized Formulation Inhaled Dose — Administered via Nebulizer
  Arms: Nebulized Formulation Inhaled Dose

SUMMARY:
This protocol will seek to enroll up to 60 immunocompromised subjects diagnosed with parainfluenza infection.

All subjects will have additional PK and Immunogenicity blood samples collected.

DETAILED DESCRIPTION:
The study will investigate the safety, tolerability, clinical and virologic effect of DAS1814 for the treatment of PIV infections in up to 60 immunocompromised patients with no other treatment options.

Eligible immunocompromised patients positively diagnosed with PIV infection will receive DAS181 by DPI or Nebulized formulation.

DPI: 10 mg DAS181 will be administered for seven (7) consecutive days for up to a total cumulative dose of 70mg.

Nebulized: DAS181 F02 formulation in solution will be administered for seven (7) consecutive days for up to a total cumulative dose of 28.9 mg.

Assessment of viral shedding and viral resistance testing will be performed on collected viral load samples. Blood samples will be obtained to evaluate safety at each scheduled visit.

Routine safety monitoring (including Adverse Event (AE) reporting, clinical laboratory tests, vital signs, electrocardiogram (ECG) and )2 levels) will be conducted in all subjects. A final safety assessment will occur at Day 28 (+/- 2 days) after enrollment/first dose of study drug. Survival, diary cards, and quality of life will be collected at Day 60 and 90. PK will be collected at each visit on all subjects from baseline/visit 2 to visit 11/Day 28. Immunogenicity samples will be collected at selected time points in all subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥12 years
2. Able to provide informed consent or child assent with parental consent
3. Immunocompromised, as defined by one of the following:

   * Allogeneic hematopoietic cell transplantation (HCT)
   * Lung or lung-heart transplantation
   * Patients treated with chemotherapy for hematologic malignancies or autologous HCT
4. Confirmed Parainfluenza virus by nasopharyngeal swab or tracheal aspirate for one of the following:

   * Respiratory virus panel
   * DFA
   * Qualitative/quantitative RT-PCR test for parainfluenza virus performed at the local laboratory (a confirmatory PCR test will be done at the central lab but is not required to start the patient on study).
5. Female subjects of child-bearing potential who are capable of conception must be:

   post-menopausal (one year or greater without menses), surgically incapable of childbearing, or practicing two effective methods of birth control. Acceptable methods include intrauterine device, spermicide, barrier, male partner surgical sterilization and hormonal contraception. A female subject must agree to practice two acceptable methods of birth control during the 28 day study period. Abstinence is not an acceptable method of contraception. All reproductive female subjects must have a negative serum pregnancy test during the screening visit.
6. Male subjects must agree to use medically accepted form of contraception during the 28 day study period.

Exclusion Criteria:

1. Psychiatric or cognitive illness or recreational drug/alcohol use that, in the opinion of the principal investigator, would affect patient safety and/or compliance.
2. Any significant finding in the patient's medical history or physical examination that, in the opinion of the investigator, would affect patient safety, ability to use the dry powder inhaler or compliance with the dosing schedule.
3. Subjects currently treated with oral, aerosolized or IV ribavirin
4. Subjects taking any investigational drug used to research or treat PIV

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-08; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence and severity of AEs, SAEs, and lab abnormalities as a measure of safety and tolerability. | 2 years

SECONDARY OUTCOMES:
Proportion of subjects with PIV viral load reduction at Day 28 | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ron Moss, MD, CEO, Study Chair — Ansun Biopharma, Inc.
Locations (23):
- United States (23):
  - City of Hope, Duarte, California
  - Children's Hospital of Orange County, Orange, California
  - Stanford University Medical Center, Palo Alto, California
  - University of Chicago, Chicago, Illinois
  - Indiana Blood and Marrow Transplantation, Indianapolis, Indiana
  - University of Kansas Cancer Center, Kansas City, Kansas
  - John Hopkins University School of Medicine, Baltimore, Maryland
  - Brigham & Women's Hospital, Boston, Massachusetts
  - University of Minnesota, School of Medicine, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Weill Cornell Medical College/New York Presbyterian Hospital, New York, New York
  - Weill Cornell Medical College-Peds, New York, New York
  - Duke University, Durham, North Carolina
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - Fred Hutchinson Cencer Research Center, Seattle, Washington